CLINICAL TRIAL: NCT01340755
Title: A Pilot Study of Laparoscopy-Assisted Transanal Endoscopy Rectosigmoid Resection for Rectal Cancer
Brief Title: Laparoscopy-Assisted Transanal Endoscopy Rectosigmoid Resection for Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Patricia Sylla, Assistant Professor of Surgery, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-409
Record Dates: First submitted 2011-04-21; First posted 2011-04-25 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Adenocarcinoma of the Rectum
Keywords: Rectal cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Transanal Endoscopic Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transanal endoscopic surgery (Experimental): Laparoscopy-assisted transanal endoscopic rectosigmoid resection
  Interventions: Procedure: Transanal endoscopic surgery

INTERVENTIONS:
Procedure: Transanal endoscopic surgery — Laparoscopy-assisted transanal endoscopic rectosigmoid resection

SUMMARY:
Transanal Endoscopic Rectosigmoid Resection with Laparoscopic Assistance was developed at Massachusetts General Hospital and performed successfully to remove cancer of the lower rectum. Based on the outcomes, the research doctors believe that this investigational surgery may be as safe and effective as standard laparoscopic or open surgery performed to remove rectal cancer, may facilitate the operation and reduce the size of the abdominal incisions. In this research study, the investigators are looking to see if this investigational procedure is a safe and effective approach to remove rectal cancer of the mid and lower rectum.

DETAILED DESCRIPTION:
Subjects will have their rectal cancer removed using a technique combining surgery through the anus and standard laparoscopy. At the end of the procedure, the rectum will be removed though the anus, the bowel will be re-connected to the anus, and a temporary diverting stoma will be created, which is standard of care following surgery for this type of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven adenocarcinoma of the rectum
* Eligible to undergo standard open or laparoscopic low anterior resection with a temporary diverting stoma
* Node negative (N0), T1 (high risk features), T2 and T3 rectal cancer on pelvic MRI
* Closest distance between tumor edge and mesorectal fascia 5mm or more based on pelvic MRI
* Rectal cancer located 4-12 cm from the anal verge
* ECOG performance status 2 or less

Exclusion Criteria:

* Metastasis
* Obstructing rectal cancer
* Synchronous colon cancer
* T3 rectal cancer not treated preoperatively with full-course chemoradiation
* Pregnant or breast-feeding
* Receiving any other study agents
* Fecal incontinence
* History of prior colorectal cancer
* History of inflammatory bowel disease
* History of pelvic radiation
* Prior pelvic surgery or multiple abdominal procedures
* BMI > 30
* Large uterine fibroids
* Uncontrolled intercurrent illness
* Other malignancies diagnosed within the previous year, except basal cell cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-03; Primary Completion 2012-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Adequacy of the total mesorectal excision based on standard guidelines on pathologic evaluation of TME specimens. | 1-5 years

SECONDARY OUTCOMES:
Incidence of 30-day perioperative complications including intraoperative, surgical postoperative, and medical postoperative complications. | 1-5 years
Incidence of long-term complications | 1-5 years
Oncologic outcomes in subjects receiving transanal endoscopic rectosigmoid resection | 1-5 years

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Sylla, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sylla P, Bordeianou LG, Berger D, Han KS, Lauwers GY, Sahani DV, Sbeih MA, Lacy AM, Rattner DW. A pilot study of natural orifice transanal endoscopic total mesorectal excision with laparoscopic assistance for rectal cancer. Surg Endosc. 2013 Sep;27(9):3396-405. doi: 10.1007/s00464-013-2922-7. Epub 2013 Apr 10. PMID 23572214